CLINICAL TRIAL: NCT01795040
Title: Efficacy of a Supplementary Balanced Diet With Omega-3/ Omega-6 Fatty Acids Among 3-6 Year Olds With Symptoms of ADHD
Brief Title: Efficacy of Omega-3/Omega-6 Fatty Acids in Pre-school Children at Risk for ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Prof. Dr., University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OMEGA-Study
Record Dates: First submitted 2013-02-16; First posted 2013-02-20 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Children With ADHD Symptoms >90th Percentile (FBB-ADHS-V); no Beginning or Completion of Psychotherapeutically or Psychopharmalogical Treatment During the Study
Keywords: omega-3/omega-6 fatty acids; Pre-school children with ADHD symptoms; randomized controlled trial
MeSH Terms: interventions — Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega-3/omega-6 fatty acids (PUFAs) (Experimental): Equazen 500mg/day= 116 mg docosahexaenoic acid, 372 mg Eicosapentaenoic acid, 40 mg gamma-Linolenic acid
  Interventions: Dietary Supplement: omega-3/omega-6 fatty acids (PUFAs)
- placebo without PUFAs (Placebo Comparator): Placebo without PUFAs
  Interventions: Dietary Supplement: omega-3/omega-6 fatty acids (PUFAs)

INTERVENTIONS:
Dietary Supplement: omega-3/omega-6 fatty acids (PUFAs) — Equazen 500mg/day= 116 mg docosahexaenoic acid, 372 mg Eicosapentaenoic acid, 40 mg gamma-Linolenic acid
  Other Names: Equazen Eye Q

SUMMARY:
The efficacy of PUFAs (as nutritional supplement) in/for pre-school children with ADHS symptoms will be evaluated in a randomised controlled doubleblind trail with children aged 3-6 years.

DETAILED DESCRIPTION:
The study aims at the reduction of hyperactivity, inattention and impulsivity in pre-school children aged 3-6 years, visiting a preschool, and the prevention of clinical ADHD symptoms. The 3-6 years old children will be identified by a combined parent and teacher rating ADHD-symptoms questionnaire (FBB-ADHS-V). Children with ADHD symptoms >90th percentile will participate in a following diagnostic process. The children (n = 150) will be randomised doubleblind to a control group (taking every day four capsules Equazen eye q, containing 400 mg fish oil and 100mg evening primrose oil - EPA (372mg), DHA (116mg), GLA (40mg) and vitamin E (7.2 mg) ) or placebo group. The study is divided into two phases with four months each. After unblinding after the first phase pre-school children taking placebo receive Omega-3/Omega-6 Fatty Acids. Children (n = 75) taking verum during first four months will be randomised doubleblind to verum or placebo. In this way the progress of the behaviour symptoms will be evaluated after a significant period of time (eigth months). Clinical examination (questionnaires, intelligence test, medical examination) and evaluation of ADHD symptoms through parents and teachers with several questionnaires will be used before beginning, after four months and after eight months. In addition the pre-school children will be taken a blood sample (finger prick test) to measure the omega-3/omega-6 fatty acids levels. Additionally regular phone calls will be implemented. Medical examinations and meetings will taken place if required. If symptoms increase, children will be treated medical and/ or psychotherapeutically.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 - 6 years
* Visit of a preschool (Kindergarten)
* Parents have a command of the German language
* Screening score >90th percentile in a combined parent and teacher screening questionnaire

Exclusion Criteria:

* Hypersensitivity or inability to components of the study product (fish oil, primrose oil, natural strawberry flavouring, bovine gelatine)
* Consumption of omega fatty acids preparation
* Consumption of fish oil-capsules

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom Checklist for pre-school children with ADHD symptoms (FBB-ADHS-V) total score rated by parents and teachers | Change from pre- assessment to post assessment four months after treatment begin and to post assessment eight months after treatment begin
  The FBB-ADHS-V Questionnaire is a developed parent and teacher rating scale which assesses several factors of hyperactivity, impulsivity and inattention problems in pre-school or at home.

SECONDARY OUTCOMES:
Change in ODD symptoms -parent/ teacher rated (FBB-ADHD-V) | Change from pre- assessment to post assessment four months after treatment begin and to post assessment eight months after treatment begin
Change in Child Behavior Checklist (CBCL) and Teacher Report Form (TRF) | Change from pre- assessment to post assessment four months after treatment begin.
  The CBCL and the TRF are well evaluated rating scales for the assessement of a broad spectrum of child behavioral and emotional problems as perceived by parents and teachers respectively
Diagnostic checklist for ADHD (DCL-ADHS) and diagnostic checklist for odd (DCL-SSV) | Change from pre- assessment to post assessment four months after treatment begin and to post assessment eight months after treatment begin
  The DCL-ADHD and the DCL-ODD are external assessment questionnaires. Parents were asked 18 questions to hyperactivity, impulsivity and inattention by the rater or to symptom criteria for ODD.
Change in intelligence: Sequential & Simultaneous Processing, Achievement (K-ABC) | Change from pre- assessment to post assessment four months after treatment begin.
  The Kaufman Assessment Battery for Children (K-ABC) is a standardized test that assesses intelligence and achievement in children aged 2;6 to 12;6 years. It is comprised of four global test scores that include: sequential processing scales, simultaneous processing scales, achievement scales and mental processing composite. There is an additional nonverbal scale.

OTHER OUTCOMES:
finger prick test to measure the PUFA blood concentration | Change from pre- assessment to post assessment four months after treatment begin
  It will taken a blood sample (finger prick test) to measure the omega-3/omega-6 fatty acids levels.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Doepfner, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry Univ. Cologne
Locations (1):
- Department of Child and Adolescent Psychiatry at the University Cologne, Cologne, Germany

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600